CLINICAL TRIAL: NCT04177394
Title: A Post-Market Study Assessment of the Safety and Performance of the MitraClip G4 System
Brief Title: MitraClip EXPAND G4 Study
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10320
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Mitral Valve Regurgitation; Mitral Regurgitation
Keywords: MitraClip; MitraClip G4; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- MitraClip G4 System: Percutaneous mitral valve repair using the MitraClip G4 system
  Interventions: Device: MitraClip G4 System

INTERVENTIONS:
Device: MitraClip G4 System — Percutaneous mitral valve repair using the MitraClip G4 system.

SUMMARY:
This primary objective of the EXPAND G4 study is to confirm the safety and performance of the MitraClip G4 System in a post-market setting.

DETAILED DESCRIPTION:
This is a post-market, multi-center, single-arm, prospective study to assess the safety and performance of the next generation MitraClip G4 System. The current protocol describes the design of this post-market study.

Up to 1,100 post-market, consented patients will be treated with a MitraClip G4 device according to local guidelines and IFU from the Europe and Middle East, the United States, Canada and Japan, and will be included in the analysis for the MitraClip EXPAND G4 Study. Follow-up echocardiograms will be collected at Discharge, 30 days and 1 year and 5 year at post-procedure visits. Additional clinical follow-up visits will be at 6 months (phone call), 2, 3, 4 year (office visits). Cardiovascular adverse events will be reported through 5 years to confirm safety of the MitraClip G4 System.

During the Phase 1 of the study 100 subjects were enrolled at 15 sites in the United States with the goal of evaluating the early safety and procedural outcomes associated with the MitraClip G4. The follow up duration was 30 days. Phase I was completed August 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled to receive the MitraClip per the current approved indications for use
2. Subjects who give consent for their participation

Exclusion Criteria:

1. Subjects participating in another clinical study that may impact the follow-up or results of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include an analysis of all consented subjects who satisfy the inclusion and exclusion criteria and who are treated with the MitraClip G4 System. The study will include approximately 1100 subjects treated with the MitraClip G4 System that have data available for assessment of APS.
Sampling Method: Probability Sample
Enrollment: 1164 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2028-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Sundareswaran, PhD, Study Director — Abbott Structural Heart
Locations (63):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cardiology Associates of Mobile, Inc., Mobile, Alabama
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Scripps Health, La Jolla, California
  - University of California - Davis Medical Center, Sacramento, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Cardiology Associates of Fairfield County, PC, Norwalk, Connecticut
  - NCH Healthcare System, Naples, Florida
  - Northshore University Health System, Evanston, Illinois
  - Prairie Education & Research, Springfield, Illinois
  - Via Christi, Wichita, Kansas
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Albany Medical Center, Albany, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Hudson Valley Cardiovascular Practice, P.C., Poughkeepsie, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - St. Thomas Hospital, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
- France (2):
  - CHU Hospital de Pontchaillou, Rennes
  - CHU Rangueil Toulouse, Toulouse
- Germany (17):
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Kiel
  - Elisabeth-Krankenhaus Essen GmbH, Essen, North Rhin
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universitat Mainz, Mainz, Rhinela
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden, Saxony
  - Universitätsklinikum Freiburg, Bad Krozingen
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen
  - Immanuelklinikum Bernau und Herzzentrum Brandenburg, Bernau
  - Medizinische Einrichtungen der Universitat zu Koln, Cologne
  - St.-Johannes-Hospital, Dortmund
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf
  - Klinikum der Justus-Liebig-Universität, Giessen
  - Universitatsmedizin Gottingen, Göttingen
  - Katholisches Marienkrankenhaus GmbH, Hamburg
  - Klinikum der Ruprecht-Karls-Universität Heidelberg, Heidelberg
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitatsklinikum Ulm, Ulm
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (4):
  - Ospedale San Raffaele- Cardiac, Milan, Lombard
  - Policlinico San Donato, Milan, Lombard
  - Presidio Ospedaliero Ferrarotto Alessi, Catania
  - Centro Cardiologico Monzino, Milan
- Japan (8):
  - Nagoya Heart Center, Nagoya, Aichi-ken
  - Gifu Prefectural General Medical Center, Gifu, Gifu
  - Hyogo Brain & Heart Center, Himeji, Hyōgo
  - Mitsui Memorial Hospital, Tokyo, Kanto
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Sendai Kosei Hospital, Sendai, Miyagi
  - The Sakakibara Heart Insitute of Okayama, Okayama, Okayama-ken
  - Toyama University Hospital, Toyama
- Erasmus Mc Rotterdam, Rotterdam, Netherlands
- Prince Sultan Cardiac Center - Riyadh, Riyadh, Saudi Arabia
- Spain (2):
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Alvaro Cunqueiro Dept of Interventional Cardiology, Vigo

REFERENCES:
- [Derived] Tang GHL, Price MJ, Rottbauer W, Mahoney PD, Hausleiter J, Raake PW, Rollefson WA, Lurz P, Denti P, Chehab BK, Dong M, Huang R, Asch FM, Zamorano JL, von Bardeleben RS, Maisano F, Kar S, Rodriguez E. Transcatheter Edge-to-Edge Repair in Secondary Mitral Regurgitation With Extended Non-COAPT-Like Features: From the EXPANDed Studies. JACC Heart Fail. 2025 Sep;13(9):102565. doi: 10.1016/j.jchf.2025.102565. Epub 2025 Jun 27. PMID 40713981
- [Derived] Morikawa T, Enta Y, Sakamoto T, Yamamoto M, Ueno H, Yagasaki H, Asch FM, Dong M, Peterman K, Rodriguez E, von Bardeleben RS, Asami M. 1-Year Outcomes of Fourth-Generation Mitral Transcatheter Edge-to-Edge Repair in Japan From the EXPAND G4 Study. JACC Asia. 2024 Sep 24;4(11):810-821. doi: 10.1016/j.jacasi.2024.08.003. eCollection 2024 Nov. PMID 39619400
- [Derived] von Bardeleben RS, Mahoney P, Morse MA, Price MJ, Denti P, Maisano F, Rogers JH, Rinaldi M, De Marco F, Rollefson W, Chehab B, Williams M, Leurent G, Asch FM, Rodriguez E. 1-Year Outcomes With Fourth-Generation Mitral Valve Transcatheter Edge-to-Edge Repair From the EXPAND G4 Study. JACC Cardiovasc Interv. 2023 Nov 13;16(21):2600-2610. doi: 10.1016/j.jcin.2023.09.029. Epub 2023 Oct 24. PMID 37877913

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MitraClip G4 System
Started | 1164
Completed (Participant Flow is for 30 Days) | 1053
Not Completed | 111
Not completed — Death | 16
Not completed — Withdrawal by Subject | 19
Not completed — Missed visits | 61
Not completed — Expected Visits | 15

BASELINE CHARACTERISTICS:
Population: All 1164 subjects completed the Baseline visit
Arm/Group | MitraClip G4 System
Number analyzed (Participants) | 1164
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 514
  Male | 650
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 3
  Canada | 7
  Netherlands | 13
  United States | 586
  Japan | 95
  Italy | 144
  Israel | 10
  France | 52
  Germany | 232
  Spain | 22
Height [Mean (Standard Deviation); unit: cm] — Population: All available data has been reported.
  cm
    number analyzed (Participants) | 1163
    (all) | 167.78 (11.26)
Weight [Mean (Standard Deviation); unit: Kg] | 73.25 (18.91)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: All available data has been reported
  kg/m^2
    number analyzed (Participants) | 1163
    (all) | 25.91 (5.89)
Euro Score II [Mean (Standard Deviation); unit: points on a scale] — EuroSCORE II estimates the 30-day mortality risk after cardiac surgery, expressed as a percentage. EuroSCORE II score has three groups, 1. low risk defined as EuroSCORE < 4%, 2. intermediate risk as 4-8%, and 3. high risk as > 8%. Population: All available data has been reported
  points on a scale
    number analyzed (Participants) | 472
    (all) | 6.48 (6.85)
STS Replacement Score [Mean (Standard Deviation); unit: percentage] — The Society of Thoracic Surgeons (STS) score is a validated risk-prediction model for open surgery based on data from the STS National Adult Cardiac Surgery Database. In general, an STS predicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% or greater is considered high risk. As of November 15, 2018, The STS released an updated short-term risk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator allows you to calculate a patient's risk of mortality and morbidities for the most commonly performed cardiac surgeries. Population: All available data has been reported
  percentage
    number analyzed (Participants) | 608
    (all) | 7.55 (6.21)
Prior Cardiac Sugeries [Count of Participants; unit: Participants] | 266
Prior Coronary Revascularization [Count of Participants; unit: Participants] | 448
Coronary Artery Bypass Graft (CABG) [Count of Participants; unit: Participants] | 176
Prior Cardiac Interventions (PCI) [Count of Participants; unit: Participants] | 364
Permanent Pacemaker [Count of Participants; unit: Participants] | 315
Prior Heart Failure Hospitalization within 1 year [Count of Participants; unit: Participants] | 472

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mitral Valve Regurgitation Severity ≤2+ at 30 Days
Description: Mitral Valve Regurgitation (MR) Severity of 2+ or less at 30 days
Time Frame: At 30 days
Population: All available data has been reported
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip G4 System
Number analyzed (Participants) | 983
Participants
  0+:None | 350
  1+: Mild | 547
  2+: Moderate | 65
  3+: Moderate to Severe | 17
  4+: Severe | 4

2. Primary Outcome: Occurrence of Major Adverse Events (MAE) at 30 Days
Description: MAE is defined as a composite of all-cause Death, Myocardial Infarction, Stroke, or non-elective Cardiovascular (CV) surgery for device related complications.
Time Frame: At 30 days
Population: All available data has been reported
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip G4 System
Number analyzed (Participants) | 1159
Participants
  All Cause Death | 16
  Myocardial Infarction | 2
  Stroke | 6
  Non-elective CV Surgery for device related complications | 10

3. Other Pre Specified Outcome: Number of Participants With APS
Description: Acute Procedural Success (APS) defined as successful implantation of the MitraClip device with resulting MR severity of 2+ or less on discharge echocardiogram. Echocardiogram (30-day echocardiogram will be used if discharge is unavailable or uninterpretable). Subjects who die or undergo mitral valve surgery before discharge are considered to be an APS failure
Time Frame: Up to 10 Days
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip G4 System
Number analyzed (Participants) | 1159
Participants | 1119

4. Other Pre Specified Outcome: Number of Participants With ADS
Description: Acute Device Success defined as successful implant of the MitraClip device without the occurrence of a Device-Related Complication (including device embolization, Single Leaflet Device Attachment (SLDA), bleeding, or perforation) through discharge.
Time Frame: Up to 10 Days
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip G4 System
Number analyzed (Participants) | 1164
Participants | 1118

5. Other Pre Specified Outcome: Occurrence of In-hospital Major Adverse Events (MAE)
Description: In-hospital Major Adverse Events (MAE) defined as the number of MAEs that occur prior to discharge from hospitalization in which MitraClip Procedure was performed.
Time Frame: Through time the subject is discharged from the hospital post-procedure, the average time ranges between 1-6 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip G4 System
Number analyzed (Participants) | 1164
Participants
  All Cause Death | 9
  Myocardial Infarction | 0
  Stroke | 3
  Non-elective CV surgery for device related complications | 9

6. Other Pre Specified Outcome: Rate of All Cause Mortality Through 5 Years
Description: All Cause Mortality Through 5 years
Time Frame: Through 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Number of Heart Failure Hospitalization Through 5 Years
Description: Heart Failure Hospitalization through 5 years
Time Frame: Through 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Occurrence of MAE
Description: Occurrence of Major Adverse Events (MAE) as defined in the protocol through 5 years
Time Frame: Through 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Rate of Device Related Complications as Defined in the Protocol Through 5 Years
Description: Device Related Complications as defined in the protocol through 5 years
Time Frame: Through 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Percentage of Participants With MR Reduction to ≤2+ or Less at Discharge, 30 Days, 1 and 5 Year
Description: MR Reduction to ≤2+ at Discharge, 30 days, 1 and 5 year
Time Frame: Through time the subject is discharged from the hospital post-procedure, the average time ranges between 1-6 days, and at 30 days, 1 and 5 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Percentage of Participants With MR Reduction to ≤1+ or Less at Discharge, 30 Days, 1 and 5 Year
Description: MR Reduction to ≤1+ at Discharge, 30 days, 1 and 5 year
Time Frame: as for outcome 10
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Difference Between New York Heart Association (NYHA) at Discharge, 30 Days, 1, 2, 3, 4 and 5 Years, Higher Class Means a Worse Outcome (Class I to IV)
Description: Difference Between NYHA Class at Discharge, 30 days, 1, 2, 3, 4 and 5 years
Time Frame: Through time the subject is discharged from the hospital post-procedure, the average time ranges between 1-6 days, and at 30 days, 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Difference Between Kansas City Cardiomyopathy Questionnaire (KCCQ) Score at 30 Days, 1, 2, 3, 4 and 5 Year, Higher Score Means a Better Outcome (0-100)
Description: Difference Between QOL at 30 days, 1, 2, 3, 4 and 5 year
Time Frame: 30 days, 1, 2, 3, 4 and 5 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Difference Between 6 Minutes Walk Distance (6MWD) at 30 Days, 1 and 5 Year
Description: Difference Between 6MWD at 30 days, 1, 2, 3, 4 and 5 year
Time Frame: 30 days, 1, 2, 3, 4 and 5 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events are reported through 30 days.
Description: Rates are reported as number of patients with an event out of the total number of patients in the study.
Arm/Group | MitraClip G4 System
All-Cause Mortality (participants affected / at risk) | 16/1164
Serious Adverse Events (participants affected / at risk) | 209/1164
Other Adverse Events (participants affected / at risk) | 0/1164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip G4 System (N=1164)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4)
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 16 (16)
ATRIAL FIBRILLATION (Cardiac disorders) | 16 (16)
ATRIAL SEPTAL DEFECT ACQUIRED (Cardiac disorders) | 8 (8)
CARDIAC FAILURE (Cardiac disorders) | 37 (37)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 16 (18)
CARDIAC PERFORATION (Cardiac disorders) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 (3)
CARDIOGENIC SHOCK (Cardiac disorders) | 14 (14)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1)
MITRAL PERFORATION (Cardiac disorders) | 9 (9)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 14 (15)
MITRAL VALVE STENOSIS (Cardiac disorders) | 3 (3)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 3 (3)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
ASTHENIA (Gastrointestinal disorders) | 2 (2)
CARDIAC COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 3 (3)
CHEST PAIN (General disorders) | 3 (3)
DEATH (General disorders) | 2 (2)
DEVICE CAPTURING ISSUE (General disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
CARDIAC INFECTION (Infections and infestations) | 3 (3)
INFECTION (Infections and infestations) | 20 (21)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 1 (1)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 9 (9)
VASCULAR PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 3 (3)
ANTICOAGULATION DRUG LEVEL BELOW THERAPEUTIC (Investigations) | 1 (1)
MEAN ARTERIAL PRESSURE DECREASED (Investigations) | 1 (1)
OXYGEN SATURATION DECREASED (Investigations) | 2 (2)
METABOLISM AND NUTRITION DISORDERS (Investigations) | 2 (2)
HYPERKALAEMIA (Investigations) | 1 (1)
METABOLIC ACIDOSIS (Investigations) | 1 (1)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 2 (2)
ISCHAEMIC STROKE (Nervous system disorders) | 5 (5)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
SIMPLE PARTIAL SEIZURES (Nervous system disorders) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1)
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 1 (1)
DELIRIUM (Psychiatric disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 18 (18)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (5)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 (4)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1)
EMBOLISM (Vascular disorders) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 39 (42)
HYPERTENSION (Vascular disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 11 (11)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT04177394/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT04177394/SAP_001.pdf